CLINICAL TRIAL: NCT06020222
Title: The Effect of Cryotherapy on Breast Cancer Patients in Kaohsiung Medical University Hospital
Brief Title: The Effect of Cryotherapy on Breast Cancer Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Collaborators: Taiwan Nurses Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: KMUHIRB-F(I)-20230041; TWNA-1121020 (Other Grant/Funding Number: Funder)
Record Dates: First submitted 2023-05-02; First posted 2023-08-31 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-05

CONDITIONS: Chemotherapy-induced Peripheral Neuropathy
Keywords: breast cancer; chemotherapy; neuropathy; cryotherapy
MeSH Terms: conditions — Breast Neoplasms | interventions — Cryotherapy; Educational Status

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Assessors don't know groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cryotherapy group (Experimental): Both hands and feet received cryotherapy gloves and boots
  Interventions: Device: cryotherapy
- Usual care group (Placebo Comparator): health education leaflets
  Interventions: Other: education

INTERVENTIONS:
Device: cryotherapy — Both hands and feet received cryotherapy gloves and boots, and the frequency was once every three weeks. Each cycle was 90 minutes, and the cycle was performed 4 times.
  Arms: Cryotherapy group
Other: education — Provide preventive CIPN education leaflets
  Arms: Usual care group

SUMMARY:
The goal of this clinical trial is to test the effect of cryotherpay on chemotherapy-induced peripheral neuropathy(CIPN) among Breast Cancer Patients. The main questions of research are:

* Does cryotherapy reduce the incidence of CIPN?
* Does cryotherapy reduce the severity of CIPN and improve the quality of life? Participants will be put on the cold gloves and boots during chemotherapy injection process and total 90 minutes.

If there is a comparison group: Researchers will compare usual care group to make sure if it effects of CIPN.

DETAILED DESCRIPTION:
This study is designed as a experiment study. In a medical center and breast ward, a randomized controlled trial was used to evaluate the effect of cryotherapy. Block sampling was adopted, and participants total 94 were included. Patients were randomly assigned to the croytherapy group (n=47) or the usual care group(n=47). Both hands and feet received cryotherapy, and the frequency was once every three weeks. Each cycle was 90-150 minutes, and the cycle was performed 4-8 times. The instrument included EPRTC QLQ-CIPN20, PNQ, and EORTC QLQ-C30. After 12-32 weeks, the cryotherapy received qualitative interviews to collect experience and perceptions. Quantitaitve data were constructed and analyzed with SPSS 20.0 version, and Chi-square test was used to detect the incidence of CIPN after three months. Mixed linear model was used to detect the severity of peripheral neuropathy symptoms and quality of life. Survival analysis was used to compare the occurrence time of peripheral neuropathy events between groups.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Breast cancer stage I-III, first time receive paclitaxel neurotoxic chemotherapy, consciousness clear, able to communicate in Taiwanese or Mandarin

Exclusion Criteria:

* Insulin depent diabetes, Raynaud's disease, cold urticaria disease, cryoglobulinemia and sclerosing basal cell carcinoma, those diagnosed with mental illness, and those with visual or hearing impairments.

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Patient neurotoxicity questionnaire (PNQ) | first day
  the incidence of sensory and motor neuropathy, the Grade A to E, the higher the grade, the more serious
Patient neurotoxicity questionnaire (PNQ) | the day after the first chemotherapy
  the incidence of sensory and motor neuropathy,the Grade A to E, the higher the grade, the more serious
Patient neurotoxicity questionnaire (PNQ) | the day after the second chemotherapy
  the incidence of sensory and motor neuropathy,the Grade A to E, the higher the grade, the more serious
Patient neurotoxicity questionnaire (PNQ) | the day after the third chemotherapy
  the incidence of sensory and motor neuropathy,the Grade A to E, the higher the grade, the more serious
Patient neurotoxicity questionnaire (PNQ) | the day after the fourth chemotherapy
  the incidence of sensory and motor neuropathy,the Grade A to E, the higher the grade, the more serious

SECONDARY OUTCOMES:
European Organization for Research and Treatment of Cancer quality of life questionnaire-chemotherapy-induced peripheral neuropathy 20 | first day
  the severity of Chemotherapy-induced peripheral neuropathy (CIPN), the higher score, the more severe
European Organization for Research and Treatment of Cancer quality of life questionnaire-chemotherapy-induced peripheral neuropathy 20 | the day after the first chemotherapy
  the severity of Chemotherapy-induced peripheral neuropathy (CIPN), the higher score, the more severe
European Organization for Research and Treatment of Cancer quality of life questionnaire-chemotherapy-induced peripheral neuropathy 20 | the day after the second chemotherapy
  the severity of Chemotherapy-induced peripheral neuropathy (CIPN), the higher score, the more severe
European Organization for Research and Treatment of Cancer quality of life questionnaire-chemotherapy-induced peripheral neuropathy 20 | the day after the third chemotherapy
  the severity of Chemotherapy-induced peripheral neuropathy (CIPN), the higher score, the more severe
European Organization for Research and Treatment of Cancer quality of life questionnaire-chemotherapy-induced peripheral neuropathy 20 | the day after the fourth chemotherapy
  the severity of Chemotherapy-induced peripheral neuropathy (CIPN), the higher score, the more severe
European Organization for the Research and Treatment of Cancer core questionnaire QLQ30 | first day
  the quality of life in breast cancer patients, higher score indicate pooer quality of life
European Organization for the Research and Treatment of Cancer core questionnaire QLQ30 | the day after the first chemotherapy
  the quality of life in breast cancer patients,higher score indicate pooer quality of life
European Organization for the Research and Treatment of Cancer core questionnaire QLQ30 | the day after the second chemotherapy
  the quality of life in breast cancer patients,higher score indicate pooer quality of life
European Organization for the Research and Treatment of Cancer core questionnaire QLQ30 | the day after the third chemotherapy
  the quality of life in breast cancer patients,higher score indicate pooer quality of life
European Organization for the Research and Treatment of Cancer core questionnaire QLQ30 | the day after the fourth chemotherapy
  the quality of life in breast cancer patients,higher score indicate pooer quality of life
TNSc(Total Neuropathy Score) | first day
  the severity of Chemotherapy-induced peripheral neuropathy (CIPN), the higher the score, the more severe the peripheal neuropathy
TNSc(Total Neuropathy Score) | the day after the first chemotherapy
  the severity of Chemotherapy-induced peripheral neuropathy (CIPN),the higher the score, the more severe the peripheal neuropathy
TNSc(Total Neuropathy Score) | the day after the second chemotherapy
  the severity of Chemotherapy-induced peripheral neuropathy (CIPN),the higher the score, the more severe the peripheal neuropathy
TNSc(Total Neuropathy Score) | the day after the third chemotherapy
  the severity of Chemotherapy-induced peripheral neuropathy (CIPN),the higher the score, the more severe the peripheal neuropathy
TNSc(Total Neuropathy Score) | the day after the fourth chemotherapy
  the severity of Chemotherapy-induced peripheral neuropathy (CIPN),the higher the score, the more severe the peripheal neuropathy

OTHER OUTCOMES:
the adverse event and discomfort | the day after the first cryotherapy
  the incidence of adverse event and discomfort during cryotherapy
the adverse event and discomfort | the day after the second cryotherapy
  the incidence of adverse event and discomfort during cryotherapy
the adverse event and discomfort | the day after the third cryotherapy
  the incidence of adverse event and discomfort during cryotherapy, the more times, the more frequent side effect
the adverse event and discomfort | the day after the fourth cryotherapy
  the incidence of adverse event and discomfort during cryotherapy,the more times, the more frequent side effect

CONTACTS AND LOCATIONS:
Overall Officials: Tsai-Rung Lin, Master, Principal Investigator — Kaohsiung Medical University
Locations (1):
- Tsai-Rung Lin, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No